CLINICAL TRIAL: NCT06314269
Title: Incidence of Perioperative Cerebrovascular Stroke in Assuit University Hospitals , Hospital Based Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohmed Alaa Eldeine Ahmed, Assistant Lecturer, Assiut University
Other Study IDs: 246810121416
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Perioperative Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perioperative cerebrovascular stroke patients: all Patients admitted to General surgery, cardiothorasic surgery and vascular surgery Depatments in assuit university hospitals during one year that will going to operation

SUMMARY:
Stroke is the most common cause of disability in elderly people (over 65years of age) and the third most common cause of death in the world . The World Health Organization estimates that one in six people globally will suffer from stroke in their lifetime.

Perioperative stroke is the most unwanted complication for patients, as well as for surgeons and anesthesiologists . The reported risk of perioperative stroke varies with the type of surgery. Its incidence is generally not high (approximate 0.1-1.9%) in non-cardiac, non-neurologic, and non-major surgery However, it may occur in up to 10% of patients undergoing high-risk cardiac or brain surgery . Patients with perioperative stroke are less likely to have a good functional outcome and have an eight-fold higher mortality compared with those without perioperative stroke

ELIGIBILITY:
Inclusion Criteria:

1. all Patients admitted to General surgery, cardiothorasic surgery and vascular surgery Depatments in assuit university hospitals during one year that will going to operation
2. ALL age Groups .
3. Both Sex.

Exclusion Criteria:

* Other surgical departments
* Patients with Syptoms that related to delayed recovery from anaesthesia .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all Patients admitted to General surgery, cardiothorasic surgery and vascular surgery Depatments in assuit university hospitals during one year that will going to operation
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
1- To determine incidence and prevalence of perioperative cerebrvosacular stroke in General surgery, cardiothorasic surgery and vascular surgery departments , Assuit university hospitalis , Egypt. | one year
  1- To determine incidence and prevalence of perioperative cerebrvosacular stroke in General surgery, cardiothorasic surgery and vascular surgery departments , Assuit university hospitalis , Egypt.

IPD SHARING:
Plan to Share IPD: Undecided